CLINICAL TRIAL: NCT03810625
Title: A Phase I, Randomized, Open Label, Two-Sequence, Two-Period Crossover Study to Evaluate the Effect of Food on the Pharmacokinetics of D-0502 Tablet in Postmenopausal Female Healthy Subjects
Brief Title: Food Effect Study of D-0502 Tablet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: InventisBio Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IBIO-302
Record Dates: First submitted 2018-12-16; First posted 2019-01-18 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Experimental): D-0502 Dose Patients will get D-0502 single agent once in the fasted state and once in the fed state.
  Interventions: Drug: D-0502
- Sequence BA (Experimental): D-0502 Dose Patients will get D-0502 single agent once in the fed state and once in the fasted state.
  Interventions: Drug: D-0502

INTERVENTIONS:
Drug: D-0502 — D-0502 oral tablets

SUMMARY:
This is an open label, randomized, balanced, single dose, two-treatment (fed vs. fasting), two-period, two-sequence crossover study of postmenopausal female healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be medically documented as healthy and acceptable at physical examination.
2. Subjects must have a BMI between 18.0 and 32.0 kg/m2 and a body weight of 45 kg or higher.
3. Subjects must have all laboratory parameters within the normal range or considered not clinically significant by the principal investigator.
4. Subjects must have a normal urinalysis, eGFR, ECG or results considered not clinically significant by the principal investigator.
5. Subjects must be female with postmenopausal status defined as meeting at least one of the following criteria:

   1. Have undergone a bilateral oophorectomy any time in life;
   2. Age ≥60 years, or
   3. Age <60 years but have cessation of regular menses ≥12 months with follicle stimulating hormone (FSH) value >40 milli-international units per milliliter (mIU/mL) and an estradiol value <40 picograms per milliliter (pg/mL) (140 picomoles per liter [pmol/L]).
6. Subjects are able to understand the study procedures and risks involved and must provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Subjects with any history or clinical manifestations of significant metabolic, hematological, pulmonary, cardiovascular, gastrointestinal, neurologic, hepatic, renal, urological or psychiatric disorders, as determined by the investigator.
2. Subjects who have any history or suspicion of kidney stones.
3. Subjects who are positive for human immunodeficiency virus (HIV), Hepatitis B, and/or Hepatitis C.
4. Subjects who have used prescription drugs, over-the-counter drugs, or natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 14 days before Day 1 of study medication dosing.
5. Subjects had undergone major surgery within 3 months prior to Day 1.
6. Subjects who is participating in a clinical research study involving the administration of an investigational or marketed drug or device, or who received any investigational test article within 5 half-lives or 30 days prior to Day 1 study medication dosing.
7. Subjects with positive urine drug screen test at screening.
8. Subjects with any condition that, in the judgment of the investigator, would place him/her at undue risk, or potentially compromise the results or interpretation of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic: area under the plasma concentration versus time curve (AUC) | Day 1 through 4, Day 7 through 11
  AUC: area under the plasma concentration versus time curve for D-0502; Unit: nM*hr
Pharmacokinetic: maximum plasma drug concentration (Cmax) | Day 1 through 4, Day 7 through 11
  Cmax: maximum plasma drug concentration of D-0502; Unit: nM
Pharmacokinetic: Time to reach the Cmax (Tmax) | Day 1 through 4, Day 7 through 11
  Tmax: Time to reach the Cmax of D-0502; Unit: hr
Pharmacokinetic: Apparent terminal half-life (t1/2) | Day 1 through 4, Day 7 through 11
  t1/2: apparent terminal half-life of D-0502; Unit: hr

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 2 weeks
  Number of treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Daytona Beach Clinical Research Unit, Daytona Beach, Florida, United States